CLINICAL TRIAL: NCT01799473
Title: A Patient Registry to Observe the Real-World Dosing and Titration of Tyvaso®
Brief Title: Tyvaso Dosing and Titration Evaluation: TyTRATE Registry
Status: Completed | Type: Observational
Sponsor: United Therapeutics (Industry)
Responsible Party: Sponsor
Other Study IDs: RIN-PH-404
Record Dates: First submitted 2013-02-12; First posted 2013-02-26 (Estimated); Last update posted 2015-03-24 (Estimated); Status verified 2014-05

CONDITIONS: Pulmonary Arterial Hypertension
Keywords: Tyvaso; PAH
MeSH Terms: conditions — Pulmonary Arterial Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No

SUMMARY:
This prospective, observational, multi-center, patient registry will follow patients who are newly initiated on Tyvaso for the treatment of Pulmonary Arterial Hypertension (PAH). Once enrolled, the patients' dose and titration will be followed for the first 6 months of treatment with Tyvaso.

A call-center will contact the patients directly at weeks 1, 2, 3, 4, 8, 12, 16, 20, and 24 to review their dose and titration schedule. In addition to patient-reported dosing data, some patient demographic information, will be collected by the investigative site at Baseline.

ELIGIBILITY:
Inclusion Criteria:

* Are newly prescribed Tyvaso for the treatment of PAH and plan to initiate therapy
* Are willing and able to be contacted by the patient call center.

Exclusion Criteria:

* Have previously received Tyvaso.
* Are currently enrolled in an interventional (non-FDA approved) PH clinical trial.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients newly initiating on Tyvaso therapy for the treatment of PAH
Sampling Method: Non-Probability Sample
Enrollment: 98 (Actual)
Dates: Start 2013-01; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Observe dose changes of Tyvaso over time | 6 Months

CONTACTS AND LOCATIONS:
Locations (52):
- United States (51):
  - The Regents of the University of California, La Jolla, California
  - UCLA Medical Center, Los Angeles, California
  - Southern California Permanente, Pasadena, California
  - Central Coast Chest Consultants, San Luis Obispo, California
  - Pacific Sleep Disorders Center, Stockton, California
  - Prime Healthcare, PC, West Hartford, Connecticut
  - Bay Area Cardiology Associates, PA, Brandon, Florida
  - Florida Lung & Sleep Specialist, Celebration, Florida
  - Jacksonville, Florida
  - Sacred Heart Medical Group, Miramar Beach, Florida
  - Cardiology Consultants, Pensacola, Florida
  - Pensacola Lung Group, Pensacola, Florida
  - Sacred Heart Medical Group, Pensacola, Florida
  - Pediatrix Cardiology Associates, Tampa, Florida
  - Doctors Hospital of Augusta, Augusta, Georgia
  - On Site Clinical Solutions, Cumming, Georgia
  - Duluth Biomedical Research, Duluth, Georgia
  - Gwinnett Consultants in Cardiology, Lawrenceville, Georgia
  - Atlanta Cardiology Consultants, Roswell, Georgia
  - Queens Medical Center - Honolulu, ‘Aiea, Hawaii
  - Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - Dor Heart and Vascular Clinic, Gurnee, Illinois
  - Loyola University of Chicago, Maywood, Illinois
  - Advocate Medical Group, Oak Brook, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - Clarian Health Methodist Hospital, Indianapolis, Indiana
  - MedStar Health Institute, Hyattsville, Maryland
  - Pulmonary and Care Associates of Baltimore, Pikesville, Maryland
  - Madison Medical Affiliates, Milwaukee, Michigan
  - Singing River Health System, Pascagoula, Mississippi
  - AZ Perfection Clinical, Union, New Jersey
  - Presbyterian Heart Group, Albuquerque, New Mexico
  - Heart and Lung Associates, PC, Bayside, New York
  - New York Methodist Hospital, Brooklyn, New York
  - Asheville Cardiology Associates, Asheville, North Carolina
  - Sanford Heart Hospital, Fargo, North Dakota
  - Children's Hospital Medical Center, Cincinnati, Ohio
  - The Cleveland Clinic Foundation, Cleveland, Ohio
  - Midwest Pulmonary & Sleep Research, Dayton, Ohio
  - Southwest General Health Center, Middleburg Heights, Ohio
  - INTEGRIS Baptist Medical Center, Inc, Oklahoma City, Oklahoma
  - The Lankenau Institute for Medical Research, Wynnewood, Pennsylvania
  - WellSpan Health, York, Pennsylvania
  - Maury Regional Medical Center, Columbia, Tennessee
  - Pulmonary Consultants of San Antonio, PA, San Antonio, Texas
  - The Rector and Visitors of the University of Virginia, Charlottesville, Virginia
  - Carilion Medical Center, Roanoke, Virginia
  - Pulmonary & Sleep Research, Spokane, Washington
  - University of Wisconsin School of Medicine and Public Health, Madison, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
  - The Medical College of Wisconsin, Inc., Milwaukee, Wisconsin
- CardioPulmonary Research Center, Guaynabo, Puerto Rico